CLINICAL TRIAL: NCT07253714
Title: THE EFFECT OF PROPRIOCEPTIVE EXERCISE TRAINING ON CERVICAL PROPRIOCEPTION, KINESIOPHOBIA, AND PAIN CATASTROPHIZING LEVELS IN SARCOPENIC GERIATRIC INDIVIDUALS RESIDING IN NURSING HOMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atılım University (Other)
Responsible Party: Principal Investigator, Beyza Doğanbaz, pyhsiotherapist, Atılım University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Beyza-ftr-02
Record Dates: First submitted 2025-01-15; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2024-12

CONDITIONS: Sarcopenia in Elderly
Keywords: sarcopenia; balance; kinesiophobia; proprioception; pain catastrophizing
MeSH Terms: conditions — Sarcopenia; Kinesiophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Cervical proprioceptive exercise and classic exercise were applied.
  Interventions: Other: Classic exercises; Other: Proprioceptive exercise training
- Control Group (Active Comparator): Classic exercise (Cervical range of motion exercise+posture exercise+isometric exercises) were applied only.
  Interventions: Other: Classic exercises

INTERVENTIONS:
Other: Classic exercises — Participants in the control group received classical exercise training for 6 weeks.
Other: Proprioceptive exercise training — Participants in the experimental group received cervical proprioception exercises in addition to classical exercise training for 6 weeks.
  Arms: Experimental group

SUMMARY:
This study investigated the effects of cervical proprioceptive exercise training on cervical proprioception, kinesiophobia and pain catastrophising in sarcopenic nursing home residents.

In this randomized controlled study, 63 nursing home residents were screened for sarcopenia based on the EWGSOP2 criteria, which include assessments of handgrip strength (Jamar dynamometer), physical performance (4-meter walking test), and muscle mass evaluated by Bioelectrical Impedance Analysis. Thirty-one residents diagnosed with sarcopenia were randomly assigned to either a control group (n = 17), which completed 12 supervised sessions of conventional exercises (postural, cervical range of motion, and isometric exercises) over six weeks, or an experimental group (n = 14), which received an additional 12 sessions of cervical proprioceptive exercises. Both groups were evaluated before and after the intervention. Cervical joint position sense, kinesiophobia, pain catastrophizing, were assessed using the Joint Position Error Test; the Tampa Scale of Kinesiophobia; the Pain Catastrophizing Scale.

ELIGIBILITY:
Inclusion criteria;

* Being 65 years of age or older,
* Being diagnosed with sarcopenia,
* Having at least 91 points or more according to the Barthel daily living activities index (being mildly dependent or completely independent),
* Having 24 points or more according to the mini mental assessment, which is considered mentally healthy.

Exclusion criteria;

* Having a disability (such as limb, vision, hearing loss),
* Having a serious neurological, orthopedic or rheumatological disorder that may affect proprioception,
* Having uncontrolled hypertension/diabetes,
* Having pain in the spine and/or extremities,
* Having a psychiatric disease diagnosis.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Assessment of cervical proprioception | 10 months
  Cervical proprioception was assessed using joint position error test. While seated, the participant faced a board positioned 90 cm away at head level, consisting of concentric circles (40 cm diameter, 1-cm increments), and wore a cap with a mounted laser pointer The participant first aligned the laser with the central point to establish the neutral position, then-with eyes open-was guided through flexion, extension, right/left rotation, and right/left lateral flexion, returning to neutral after each movement. The same six movements were then actively performed with eyes closed . Six repetitions were completed for each direction, and the point at which the laser stopped was marked on the board after every trial . The mean of these points was calculated, and angular deviation from the target was determined using the arctan method based on the fixed distance to the board. A deviation of more than 4 degrees was considered to indicate impaired proprioception.

SECONDARY OUTCOMES:
Assessment of kinesiophobia | 10 months
  Kinesiophobia was assessed using the Kinesiophobia Causes Scale (KCS) . Developed by Kocjan and Knapik (2014), the scale identifies the biological and psychological sources of fear of movement and contributes to understanding the underlying causes of reduced motor activity. It comprises two domains: biological and psychological. The biological domain includes morphological factors, movement requirements, energy resources, biological drives, negative experiences, motor competence, and beliefs related to body care, while the psychological domain assesses factors such as confidence, self-efficacy, and social interaction that contribute to avoidance behavior. The Turkish validity and reliability study was conducted by Çayır et al. (2020). The scale consists of 20 items rated on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree). Higher scores indicate greater fear of movement.
Assessment of pain catastrophizing | 10 months
  Pain catastrophizing was assessed using the Pain Catastrophizing Scale (PCS), a 13-item measure evaluating maladaptive thoughts and feelings related to pain. The scale includes three subdimensions: helplessness, magnification, and rumination . Each item is scored on a 0-4 scale, and subscale scores are obtained by summing the corresponding items; the total PCS score is calculated as the sum of all items . The Turkish validity and reliability study was conducted by Uğurlu et al. (2017) . Total scores range from 0 to 52, with higher scores indicating greater pain catastrophizing.Scores above 30 reflect clinically significant levels of catastrophizing.

CONTACTS AND LOCATIONS:
Locations (1):
- Nevia Oran Nursing Home, Ankara, çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Vincent HK, George SZ, Seay AN, Vincent KR, Hurley RW. Resistance exercise, disability, and pain catastrophizing in obese adults with back pain. Med Sci Sports Exerc. 2014 Sep;46(9):1693-701. doi: 10.1249/MSS.0000000000000294. PMID 25133997
- [Background] Hayden JA, van Tulder MW, Malmivaara A, Koes BW. Exercise therapy for treatment of non-specific low back pain. Cochrane Database Syst Rev. 2005 Jul 20;2005(3):CD000335. doi: 10.1002/14651858.CD000335.pub2. PMID 16034851
- [Background] Carter IR, Lord JL. Clinical inquiries. How effective are exercise and physical therapy for chronic low back pain? J Fam Pract. 2002 Mar;51(3):209. No abstract available. PMID 11978228
- [Background] Cruz-Diaz D, Romeu M, Velasco-Gonzalez C, Martinez-Amat A, Hita-Contreras F. The effectiveness of 12 weeks of Pilates intervention on disability, pain and kinesiophobia in patients with chronic low back pain: a randomized controlled trial. Clin Rehabil. 2018 Sep;32(9):1249-1257. doi: 10.1177/0269215518768393. Epub 2018 Apr 13. PMID 29651872
- [Background] Suzuki T, Kim H, Yoshida H, Ishizaki T. Randomized controlled trial of exercise intervention for the prevention of falls in community-dwelling elderly Japanese women. J Bone Miner Metab. 2004;22(6):602-11. doi: 10.1007/s00774-004-0530-2. PMID 15490272
- [Background] Ishak NA, Zahari Z, Justine M. Kinesiophobia, Pain, Muscle Functions, and Functional Performances among Older Persons with Low Back Pain. Pain Res Treat. 2017;2017:3489617. doi: 10.1155/2017/3489617. Epub 2017 May 29. PMID 28634547
- [Background] Mortazavi H, Tabatabaeichehr M, Golestani A, Armat MR, Yousefi MR. The Effect of Tai Chi Exercise on the Risk and Fear of Falling in Older Adults: a Randomized Clinical Trial. Mater Sociomed. 2018 Mar;30(1):38-42. doi: 10.5455/msm.2018.30.38-42. PMID 29670476
- [Background] Stubbs B, Patchay S, Soundy A, Schofield P. The avoidance of activities due to fear of falling contributes to sedentary behavior among community-dwelling older adults with chronic musculoskeletal pain: a multisite observational study. Pain Med. 2014 Nov;15(11):1861-71. doi: 10.1111/pme.12570. Epub 2014 Sep 16. PMID 25224385
- [Background] Wijlhuizen GJ, de Jong R, Hopman-Rock M. Older persons afraid of falling reduce physical activity to prevent outdoor falls. Prev Med. 2007 Mar;44(3):260-4. doi: 10.1016/j.ypmed.2006.11.003. Epub 2006 Dec 19. PMID 17184828
- [Background] Murphy SL, Williams CS, Gill TM. Characteristics associated with fear of falling and activity restriction in community-living older persons. J Am Geriatr Soc. 2002 Mar;50(3):516-20. doi: 10.1046/j.1532-5415.2002.50119.x. PMID 11943049
- [Background] Vlaeyen JWS, Kole-Snijders AMJ, Boeren RGB, van Eek H. Fear of movement/(re)injury in chronic low back pain and its relation to behavioral performance. Pain. 1995 Sep;62(3):363-372. doi: 10.1016/0304-3959(94)00279-N. PMID 8657437
- [Background] Varni JW, Burwinkle TM, Lane MM. Health-related quality of life measurement in pediatric clinical practice: an appraisal and precept for future research and application. Health Qual Life Outcomes. 2005 May 16;3:34. doi: 10.1186/1477-7525-3-34. PMID 15904527
- [Background] Mohamed AA. Can Proprioceptive Training Enhance Fatigability and Decrease Progression Rate of Sarcopenia in Seniors? A Novel Approach. Curr Rheumatol Rev. 2021;17(1):58-67. doi: 10.2174/1573397116666200429113226. PMID 32348231
- [Background] Dover G, Powers ME. Reliability of Joint Position Sense and Force-Reproduction Measures During Internal and External Rotation of the Shoulder. J Athl Train. 2003 Dec;38(4):304-310. PMID 14737211
- [Background] Mustian KM, Sprod LK, Palesh OG, Peppone LJ, Janelsins MC, Mohile SG, Carroll J. Exercise for the management of side effects and quality of life among cancer survivors. Curr Sports Med Rep. 2009 Nov-Dec;8(6):325-30. doi: 10.1249/JSR.0b013e3181c22324. PMID 19904073
- [Background] Hillier S, Immink M, Thewlis D. Assessing Proprioception: A Systematic Review of Possibilities. Neurorehabil Neural Repair. 2015 Nov-Dec;29(10):933-49. doi: 10.1177/1545968315573055. Epub 2015 Feb 23. PMID 25712470
- [Background] Perez-Cabezas V, Ruiz-Molinero C, Jimenez-Rejano JJ, Chamorro-Moriana G, Gonzalez-Medina G, Chillon-Martinez R. Effectiveness of an Eye-Cervical Re-Education Program in Chronic Neck Pain: A Randomized Clinical Trial. Evid Based Complement Alternat Med. 2020 Feb 26;2020:2760413. doi: 10.1155/2020/2760413. eCollection 2020. PMID 32184889
- [Background] Pinsault N, Fleury A, Virone G, Bouvier B, Vaillant J, Vuillerme N. Test-retest reliability of cervicocephalic relocation test to neutral head position. Physiother Theory Pract. 2008 Sep-Oct;24(5):380-91. doi: 10.1080/09593980701884824. PMID 18821444
- [Background] Wannaprom N, Treleaven J, Jull G, Uthaikhup S. Neck muscle vibration produces diverse responses in balance and gait speed between individuals with and without neck pain. Musculoskelet Sci Pract. 2018 Jun;35:25-29. doi: 10.1016/j.msksp.2018.02.001. Epub 2018 Feb 5. PMID 29427867
- [Background] Corneil BD, Olivier E, Munoz DP. Neck muscle responses to stimulation of monkey superior colliculus. I. Topography and manipulation of stimulation parameters. J Neurophysiol. 2002 Oct;88(4):1980-99. doi: 10.1152/jn.2002.88.4.1980. PMID 12364523
- [Background] Grace Gaerlan M, Alpert PT, Cross C, Louis M, Kowalski S. Postural balance in young adults: the role of visual, vestibular and somatosensory systems. J Am Acad Nurse Pract. 2012 Jun;24(6):375-81. doi: 10.1111/j.1745-7599.2012.00699.x. Epub 2012 Mar 29. PMID 22672489
- [Background] Kulkarni V, Chandy MJ, Babu KS. Quantitative study of muscle spindles in suboccipital muscles of human foetuses. Neurol India. 2001 Dec;49(4):355-9. PMID 11799407
- [Background] Humphreys BK. Cervical outcome measures: testing for postural stability and balance. J Manipulative Physiol Ther. 2008 Sep;31(7):540-6. doi: 10.1016/j.jmpt.2008.08.007. PMID 18804005
- [Background] Luan H, Gdowski MJ, Newlands SD, Gdowski GT. Convergence of vestibular and neck proprioceptive sensory signals in the cerebellar interpositus. J Neurosci. 2013 Jan 16;33(3):1198-210a. doi: 10.1523/JNEUROSCI.3460-12.2013. PMID 23325256
- [Background] Aman JE, Elangovan N, Yeh IL, Konczak J. The effectiveness of proprioceptive training for improving motor function: a systematic review. Front Hum Neurosci. 2015 Jan 28;8:1075. doi: 10.3389/fnhum.2014.01075. eCollection 2014. PMID 25674059
- [Background] Ghez C, Gordon J, Ghilardi MF. Impairments of reaching movements in patients without proprioception. II. Effects of visual information on accuracy. J Neurophysiol. 1995 Jan;73(1):361-72. doi: 10.1152/jn.1995.73.1.361. PMID 7714578
- [Background] Tinetti ME, Speechley M, Ginter SF. Risk factors for falls among elderly persons living in the community. N Engl J Med. 1988 Dec 29;319(26):1701-7. doi: 10.1056/NEJM198812293192604. PMID 3205267
- [Background] Woollacott MH, Shumway-Cook A, Nashner LM. Aging and posture control: changes in sensory organization and muscular coordination. Int J Aging Hum Dev. 1986;23(2):97-114. doi: 10.2190/VXN3-N3RT-54JB-X16X. PMID 3557634
- [Background] Ferlinc A, Fabiani E, Velnar T, Gradisnik L. The Importance and Role of Proprioception in the Elderly: a Short Review. Mater Sociomed. 2019 Sep;31(3):219-221. doi: 10.5455/msm.2019.31.219-221. PMID 31762707
- [Background] Martinez-Amat A, Hita-Contreras F, Lomas-Vega R, Caballero-Martinez I, Alvarez PJ, Martinez-Lopez E. Effects of 12-week proprioception training program on postural stability, gait, and balance in older adults: a controlled clinical trial. J Strength Cond Res. 2013 Aug;27(8):2180-8. doi: 10.1519/JSC.0b013e31827da35f. PMID 23207891
- [Background] Concha-Cisternas Y, Castro-Pinero J, Leiva-Ordonez AM, Valdes-Badilla P, Celis-Morales C, Guzman-Munoz E. Effects of Neuromuscular Training on Physical Performance in Older People: A Systematic Review. Life (Basel). 2023 Mar 24;13(4):869. doi: 10.3390/life13040869. PMID 37109398
- [Background] Ager AL, Borms D, Deschepper L, Dhooghe R, Dijkhuis J, Roy JS, Cools A. Proprioception: How is it affected by shoulder pain? A systematic review. J Hand Ther. 2020 Oct-Dec;33(4):507-516. doi: 10.1016/j.jht.2019.06.002. Epub 2019 Aug 31. PMID 31481340
- [Background] Kirk B, Zanker J, Bani Hassan E, Bird S, Brennan-Olsen S, Duque G. Sarcopenia Definitions and Outcomes Consortium (SDOC) Criteria are Strongly Associated With Malnutrition, Depression, Falls, and Fractures in High-Risk Older Persons. J Am Med Dir Assoc. 2021 Apr;22(4):741-745. doi: 10.1016/j.jamda.2020.06.050. Epub 2020 Aug 6. PMID 32771358
- [Background] Kato T, Ikezoe T, Tabara Y, Matsuda F, Tsuboyama T, Ichihashi N. Differences in lower limb muscle strength and balance ability between sarcopenia stages depend on sex in community-dwelling older adults. Aging Clin Exp Res. 2022 Mar;34(3):527-534. doi: 10.1007/s40520-021-01952-6. Epub 2021 Aug 20. PMID 34417732
- [Background] Gadelha AB, Neri SGR, Oliveira RJ, Bottaro M, David AC, Vainshelboim B, Lima RM. Severity of sarcopenia is associated with postural balance and risk of falls in community-dwelling older women. Exp Aging Res. 2018 May-Jun;44(3):258-269. doi: 10.1080/0361073X.2018.1449591. Epub 2018 Mar 20. PMID 29558320
- [Background] Bohannon RW, Larkin PA, Cook AC, Gear J, Singer J. Decrease in timed balance test scores with aging. Phys Ther. 1984 Jul;64(7):1067-70. doi: 10.1093/ptj/64.7.1067. PMID 6739548
- [Background] Jacquemont S, Hagerman RJ, Hagerman PJ, Leehey MA. Fragile-X syndrome and fragile X-associated tremor/ataxia syndrome: two faces of FMR1. Lancet Neurol. 2007 Jan;6(1):45-55. doi: 10.1016/S1474-4422(06)70676-7. PMID 17166801
- [Background] Ziakas A, Klinke P, Mildenberger R, Fretz E, Williams M, Della Siega A, Kinloch D, Hilton D. Comparison of the radial and the femoral approaches in percutaneous coronary intervention for acute myocardial infarction. Am J Cardiol. 2003 Mar 1;91(5):598-600. doi: 10.1016/s0002-9149(02)03316-7. No abstract available. PMID 12615270
- [Background] Tinetti ME, McAvay G, Claus E. Does multiple risk factor reduction explain the reduction in fall rate in the Yale FICSIT Trial? Frailty and Injuries Cooperative Studies of Intervention Techniques. Am J Epidemiol. 1996 Aug 15;144(4):389-99. doi: 10.1093/oxfordjournals.aje.a008940. PMID 8712196
- [Background] Lipsitz LA, Jonsson PV, Kelley MM, Koestner JS. Causes and correlates of recurrent falls in ambulatory frail elderly. J Gerontol. 1991 Jul;46(4):M114-22. doi: 10.1093/geronj/46.4.m114. PMID 2071832
- [Background] Cuevas-Trisan R. Balance Problems and Fall Risks in the Elderly. Phys Med Rehabil Clin N Am. 2017 Nov;28(4):727-737. doi: 10.1016/j.pmr.2017.06.006. PMID 29031339
- [Background] Berger J, Bunout D, Barrera G, de la Maza MP, Henriquez S, Leiva L, Hirsch S. Rectus femoris (RF) ultrasound for the assessment of muscle mass in older people. Arch Gerontol Geriatr. 2015 Jul-Aug;61(1):33-8. doi: 10.1016/j.archger.2015.03.006. Epub 2015 Apr 1. PMID 25890633
- [Background] Lopez P, Wilhelm EN, Rech A, Minozzo F, Radaelli R, Pinto RS. Echo intensity independently predicts functionality in sedentary older men. Muscle Nerve. 2017 Jan;55(1):9-15. doi: 10.1002/mus.25168. Epub 2016 Oct 11. PMID 27145419
- [Background] Rech A, Radaelli R, Goltz FR, da Rosa LH, Schneider CD, Pinto RS. Echo intensity is negatively associated with functional capacity in older women. Age (Dordr). 2014;36(5):9708. doi: 10.1007/s11357-014-9708-2. Epub 2014 Aug 29. PMID 25167965
- [Background] Cadore EL, Izquierdo M, Conceicao M, Radaelli R, Pinto RS, Baroni BM, Vaz MA, Alberton CL, Pinto SS, Cunha G, Bottaro M, Kruel LF. Echo intensity is associated with skeletal muscle power and cardiovascular performance in elderly men. Exp Gerontol. 2012 Jun;47(6):473-8. doi: 10.1016/j.exger.2012.04.002. Epub 2012 Apr 14. PMID 22525196
- [Background] Watanabe Y, Yamada Y, Fukumoto Y, Ishihara T, Yokoyama K, Yoshida T, Miyake M, Yamagata E, Kimura M. Echo intensity obtained from ultrasonography images reflecting muscle strength in elderly men. Clin Interv Aging. 2013;8:993-8. doi: 10.2147/CIA.S47263. Epub 2013 Jul 25. PMID 23926426
- [Background] Fukumoto Y, Ikezoe T, Yamada Y, Tsukagoshi R, Nakamura M, Mori N, Kimura M, Ichihashi N. Skeletal muscle quality assessed from echo intensity is associated with muscle strength of middle-aged and elderly persons. Eur J Appl Physiol. 2012 Apr;112(4):1519-25. doi: 10.1007/s00421-011-2099-5. Epub 2011 Aug 17. PMID 21847576
- [Background] Ozcakar L, Tok F, De Muynck M, Vanderstraeten G. Musculoskeletal ultrasonography in physical and rehabilitation medicine. J Rehabil Med. 2012 Apr;44(4):310-8. doi: 10.2340/16501977-0959. PMID 22402760
- [Background] Chang KV, Wu WT, Huang KC, Jan WH, Han DS. Limb muscle quality and quantity in elderly adults with dynapenia but not sarcopenia: An ultrasound imaging study. Exp Gerontol. 2018 Jul 15;108:54-61. doi: 10.1016/j.exger.2018.03.019. Epub 2018 Mar 28. PMID 29604401
- [Background] Silva RR, Galvao LL, Meneguci J, Santos DAT, Virtuoso Junior JS, Tribess S. Dynapenia in all-cause mortality and its relationship with sedentary behavior in community-dwelling older adults. Sports Med Health Sci. 2022 Sep 23;4(4):253-259. doi: 10.1016/j.smhs.2022.09.002. eCollection 2022 Dec. PMID 36600974
- [Background] Ates Bulut E, Soysal P, Aydin AE, Dokuzlar O, Kocyigit SE, Isik AT. Vitamin B12 deficiency might be related to sarcopenia in older adults. Exp Gerontol. 2017 Sep;95:136-140. doi: 10.1016/j.exger.2017.05.017. Epub 2017 May 23. PMID 28549839
- [Background] Alexandre Tda S, Duarte YA, Santos JL, Wong R, Lebrao ML. Sarcopenia according to the European Working Group on Sarcopenia in Older People (EWGSOP) versus dynapenia as a risk factor for mortality in the elderly. J Nutr Health Aging. 2014;18(8):751-6. doi: 10.1007/s12603-014-0540-2. PMID 25286455
- [Background] Joosten E, Detroyer E, Milisen K. Effect of anaemia on hand grip strength, walking speed, functionality and 1 year mortality in older hospitalized patients. BMC Geriatr. 2016 Aug 19;16(1):153. doi: 10.1186/s12877-016-0326-y. PMID 27543049
- [Background] Reijnierse EM, de Jong N, Trappenburg MC, Blauw GJ, Butler-Browne G, Gapeyeva H, Hogrel JY, McPhee JS, Narici MV, Sipila S, Stenroth L, van Lummel RC, Pijnappels M, Meskers CGM, Maier AB. Assessment of maximal handgrip strength: how many attempts are needed? J Cachexia Sarcopenia Muscle. 2017 Jun;8(3):466-474. doi: 10.1002/jcsm.12181. Epub 2017 Feb 2. PMID 28150387
- [Background] Matteini AM, Tanaka T, Karasik D, Atzmon G, Chou WC, Eicher JD, Johnson AD, Arnold AM, Callisaya ML, Davies G, Evans DS, Holtfreter B, Lohman K, Lunetta KL, Mangino M, Smith AV, Smith JA, Teumer A, Yu L, Arking DE, Buchman AS, Chibinik LB, De Jager PL, Evans DA, Faul JD, Garcia ME, Gillham-Nasenya I, Gudnason V, Hofman A, Hsu YH, Ittermann T, Lahousse L, Liewald DC, Liu Y, Lopez L, Rivadeneira F, Rotter JI, Siggeirsdottir K, Starr JM, Thomson R, Tranah GJ, Uitterlinden AG, Volker U, Volzke H, Weir DR, Yaffe K, Zhao W, Zhuang WV, Zmuda JM, Bennett DA, Cummings SR, Deary IJ, Ferrucci L, Harris TB, Kardia SL, Kocher T, Kritchevsky SB, Psaty BM, Seshadri S, Spector TD, Srikanth VK, Windham BG, Zillikens MC, Newman AB, Walston JD, Kiel DP, Murabito JM. GWAS analysis of handgrip and lower body strength in older adults in the CHARGE consortium. Aging Cell. 2016 Oct;15(5):792-800. doi: 10.1111/acel.12468. Epub 2016 Jun 21. PMID 27325353
- [Background] Tieland M, Trouwborst I, Clark BC. Skeletal muscle performance and ageing. J Cachexia Sarcopenia Muscle. 2018 Feb;9(1):3-19. doi: 10.1002/jcsm.12238. Epub 2017 Nov 19. PMID 29151281
- [Background] Manini TM, Clark BC. Dynapenia and aging: an update. J Gerontol A Biol Sci Med Sci. 2012 Jan;67(1):28-40. doi: 10.1093/gerona/glr010. Epub 2011 Mar 28. PMID 21444359
- [Background] Iwamura M, Kanauchi M. A cross-sectional study of the association between dynapenia and higher-level functional capacity in daily living in community-dwelling older adults in Japan. BMC Geriatr. 2017 Jan 3;17(1):1. doi: 10.1186/s12877-016-0400-5. PMID 28049446
- [Background] Clark BC, Manini TM. Sarcopenia =/= dynapenia. J Gerontol A Biol Sci Med Sci. 2008 Aug;63(8):829-34. doi: 10.1093/gerona/63.8.829. PMID 18772470
- [Background] Scott D, Sanders KM, Aitken D, Hayes A, Ebeling PR, Jones G. Sarcopenic obesity and dynapenic obesity: 5-year associations with falls risk in middle-aged and older adults. Obesity (Silver Spring). 2014 Jun;22(6):1568-74. doi: 10.1002/oby.20734. Epub 2014 Mar 13. PMID 24585708
- [Background] Clark BC, Manini TM. Functional consequences of sarcopenia and dynapenia in the elderly. Curr Opin Clin Nutr Metab Care. 2010 May;13(3):271-6. doi: 10.1097/MCO.0b013e328337819e. PMID 20154609
- [Background] Scott D, Daly RM, Sanders KM, Ebeling PR. Fall and Fracture Risk in Sarcopenia and Dynapenia With and Without Obesity: the Role of Lifestyle Interventions. Curr Osteoporos Rep. 2015 Aug;13(4):235-44. doi: 10.1007/s11914-015-0274-z. PMID 26040576
- [Background] Clark BC, Manini TM. What is dynapenia? Nutrition. 2012 May;28(5):495-503. doi: 10.1016/j.nut.2011.12.002. PMID 22469110
- [Background] Sculthorpe NF, Herbert P, Grace F. One session of high-intensity interval training (HIIT) every 5 days, improves muscle power but not static balance in lifelong sedentary ageing men: A randomized controlled trial. Medicine (Baltimore). 2017 Feb;96(6):e6040. doi: 10.1097/MD.0000000000006040. PMID 28178145
- [Background] Seldeen KL, Redae YZ, Thiyagarajan R, Berman RN, Leiker MM, Troen BR. High intensity interval training improves physical performance in aged female mice: A comparison of mouse frailty assessment tools. Mech Ageing Dev. 2019 Jun;180:49-62. doi: 10.1016/j.mad.2019.04.001. Epub 2019 Apr 2. PMID 30951786
- [Background] Shen Y, Shi Q, Nong K, Li S, Yue J, Huang J, Dong B, Beauchamp M, Hao Q. Exercise for sarcopenia in older people: A systematic review and network meta-analysis. J Cachexia Sarcopenia Muscle. 2023 Jun;14(3):1199-1211. doi: 10.1002/jcsm.13225. Epub 2023 Apr 14. PMID 37057640
- [Background] Negm AM, Lee J, Hamidian R, Jones CA, Khadaroo RG. Management of Sarcopenia: A Network Meta-Analysis of Randomized Controlled Trials. J Am Med Dir Assoc. 2022 May;23(5):707-714. doi: 10.1016/j.jamda.2022.01.057. Epub 2022 Feb 18. PMID 35183490
- [Background] Yoo SZ, No MH, Heo JW, Park DH, Kang JH, Kim SH, Kwak HB. Role of exercise in age-related sarcopenia. J Exerc Rehabil. 2018 Aug 24;14(4):551-558. doi: 10.12965/jer.1836268.134. eCollection 2018 Aug. PMID 30276173
- [Background] Short KR, Vittone JL, Bigelow ML, Proctor DN, Nair KS. Age and aerobic exercise training effects on whole body and muscle protein metabolism. Am J Physiol Endocrinol Metab. 2004 Jan;286(1):E92-101. doi: 10.1152/ajpendo.00366.2003. Epub 2003 Sep 23. PMID 14506079
- [Background] Konopka AR, Harber MP. Skeletal muscle hypertrophy after aerobic exercise training. Exerc Sport Sci Rev. 2014 Apr;42(2):53-61. doi: 10.1249/JES.0000000000000007. PMID 24508740
- [Background] Beckwee D, Delaere A, Aelbrecht S, Baert V, Beaudart C, Bruyere O, de Saint-Hubert M, Bautmans I. Exercise Interventions for the Prevention and Treatment of Sarcopenia. A Systematic Umbrella Review. J Nutr Health Aging. 2019;23(6):494-502. doi: 10.1007/s12603-019-1196-8. PMID 31233069
- [Background] Chen N, He X, Feng Y, Ainsworth BE, Liu Y. Effects of resistance training in healthy older people with sarcopenia: a systematic review and meta-analysis of randomized controlled trials. Eur Rev Aging Phys Act. 2021 Nov 11;18(1):23. doi: 10.1186/s11556-021-00277-7. PMID 34763651
- [Background] Hughes VA, Roubenoff R, Wood M, Frontera WR, Evans WJ, Fiatarone Singh MA. Anthropometric assessment of 10-y changes in body composition in the elderly. Am J Clin Nutr. 2004 Aug;80(2):475-82. doi: 10.1093/ajcn/80.2.475. PMID 15277173
- [Background] Johnston AP, De Lisio M, Parise G. Resistance training, sarcopenia, and the mitochondrial theory of aging. Appl Physiol Nutr Metab. 2008 Feb;33(1):191-9. doi: 10.1139/H07-141. PMID 18347672
- [Background] Burton LA, Sumukadas D. Optimal management of sarcopenia. Clin Interv Aging. 2010 Sep 7;5:217-28. doi: 10.2147/cia.s11473. PMID 20852669
- [Background] Lacroix A, Kressig RW, Muehlbauer T, Gschwind YJ, Pfenninger B, Bruegger O, Granacher U. Effects of a Supervised versus an Unsupervised Combined Balance and Strength Training Program on Balance and Muscle Power in Healthy Older Adults: A Randomized Controlled Trial. Gerontology. 2016;62(3):275-88. doi: 10.1159/000442087. Epub 2015 Dec 9. PMID 26645282
- [Background] Marques EA, Figueiredo P, Harris TB, Wanderley FA, Carvalho J. Are resistance and aerobic exercise training equally effective at improving knee muscle strength and balance in older women? Arch Gerontol Geriatr. 2017 Jan-Feb;68:106-112. doi: 10.1016/j.archger.2016.10.002. Epub 2016 Oct 11. PMID 27764726
- [Background] Lo JH, U KP, Yiu T, Ong MT, Lee WY. Sarcopenia: Current treatments and new regenerative therapeutic approaches. J Orthop Translat. 2020 Apr 30;23:38-52. doi: 10.1016/j.jot.2020.04.002. eCollection 2020 Jul. PMID 32489859
- [Background] Rolland Y, Onder G, Morley JE, Gillette-Guyonet S, Abellan van Kan G, Vellas B. Current and future pharmacologic treatment of sarcopenia. Clin Geriatr Med. 2011 Aug;27(3):423-47. doi: 10.1016/j.cger.2011.03.008. Epub 2011 May 14. PMID 21824556
- [Background] Vestergaard S, Patel KV, Bandinelli S, Ferrucci L, Guralnik JM. Characteristics of 400-meter walk test performance and subsequent mortality in older adults. Rejuvenation Res. 2009 Jun;12(3):177-84. doi: 10.1089/rej.2009.0853. PMID 19594326
- [Background] Beaudart C, McCloskey E, Bruyere O, Cesari M, Rolland Y, Rizzoli R, Araujo de Carvalho I, Amuthavalli Thiyagarajan J, Bautmans I, Bertiere MC, Brandi ML, Al-Daghri NM, Burlet N, Cavalier E, Cerreta F, Cherubini A, Fielding R, Gielen E, Landi F, Petermans J, Reginster JY, Visser M, Kanis J, Cooper C. Sarcopenia in daily practice: assessment and management. BMC Geriatr. 2016 Oct 5;16(1):170. doi: 10.1186/s12877-016-0349-4. PMID 27716195
- [Background] Maggio M, Ceda GP, Ticinesi A, De Vita F, Gelmini G, Costantino C, Meschi T, Kressig RW, Cesari M, Fabi M, Lauretani F. Instrumental and Non-Instrumental Evaluation of 4-Meter Walking Speed in Older Individuals. PLoS One. 2016 Apr 14;11(4):e0153583. doi: 10.1371/journal.pone.0153583. eCollection 2016. PMID 27077744
- [Background] Lustgarten MS, Fielding RA. Assessment of analytical methods used to measure changes in body composition in the elderly and recommendations for their use in phase II clinical trials. J Nutr Health Aging. 2011 May;15(5):368-75. doi: 10.1007/s12603-011-0049-x. PMID 21528163
- [Background] Ashwell M, Cole TJ, Dixon AK. Obesity: new insight into the anthropometric classification of fat distribution shown by computed tomography. Br Med J (Clin Res Ed). 1985 Jun 8;290(6483):1692-4. doi: 10.1136/bmj.290.6483.1692. PMID 3924217
- [Background] Plourde G. The role of radiologic methods in assessing body composition and related metabolic parameters. Nutr Rev. 1997 Aug;55(8):289-96. doi: 10.1111/j.1753-4887.1997.tb05487.x. PMID 9287478
- [Background] Goodpaster BH, Thaete FL, Kelley DE. Composition of skeletal muscle evaluated with computed tomography. Ann N Y Acad Sci. 2000 May;904:18-24. doi: 10.1111/j.1749-6632.2000.tb06416.x. PMID 10865705
- [Background] Guerri S, Mercatelli D, Aparisi Gomez MP, Napoli A, Battista G, Guglielmi G, Bazzocchi A. Quantitative imaging techniques for the assessment of osteoporosis and sarcopenia. Quant Imaging Med Surg. 2018 Feb;8(1):60-85. doi: 10.21037/qims.2018.01.05. PMID 29541624
- [Background] Rolland Y, Czerwinski S, Abellan Van Kan G, Morley JE, Cesari M, Onder G, Woo J, Baumgartner R, Pillard F, Boirie Y, Chumlea WM, Vellas B. Sarcopenia: its assessment, etiology, pathogenesis, consequences and future perspectives. J Nutr Health Aging. 2008 Aug-Sep;12(7):433-50. doi: 10.1007/BF02982704. PMID 18615225
- [Background] McCarthy EK, Horvat MA, Holtsberg PA, Wisenbaker JM. Repeated chair stands as a measure of lower limb strength in sexagenarian women. J Gerontol A Biol Sci Med Sci. 2004 Nov;59(11):1207-12. doi: 10.1093/gerona/59.11.1207. PMID 15602077
- [Background] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Background] Yoshiko A, Ogawa M, Shimizu K, Radaelli R, Neske R, Maeda H, Maeda K, Teodoro J, Tanaka N, Pinto RS, Akima H. Chair sit-to-stand performance is associated with diagnostic features of sarcopenia in older men and women. Arch Gerontol Geriatr. 2021 Sep-Oct;96:104463. doi: 10.1016/j.archger.2021.104463. Epub 2021 Jun 14. PMID 34218157
- [Background] Testa G, Vescio A, Zuccala D, Petrantoni V, Amico M, Russo GI, Sessa G, Pavone V. Diagnosis, Treatment and Prevention of Sarcopenia in Hip Fractured Patients: Where We Are and Where We Are Going: A Systematic Review. J Clin Med. 2020 Sep 17;9(9):2997. doi: 10.3390/jcm9092997. PMID 32957453
- [Background] Carmeli E, Imam B, Merrick J. The relationship of pre-sarcopenia (low muscle mass) and sarcopenia (loss of muscle strength) with functional decline in individuals with intellectual disability (ID). Arch Gerontol Geriatr. 2012 Jul-Aug;55(1):181-5. doi: 10.1016/j.archger.2011.06.032. Epub 2011 Jul 20. PMID 21764145
- [Background] Harris-Love MO, Benson K, Leasure E, Adams B, McIntosh V. The Influence of Upper and Lower Extremity Strength on Performance-Based Sarcopenia Assessment Tests. J Funct Morphol Kinesiol. 2018 Dec;3(4):53. doi: 10.3390/jfmk3040053. Epub 2018 Nov 3. PMID 30533549
- [Background] Cruz-Jentoft AJ, Landi F, Schneider SM, Zuniga C, Arai H, Boirie Y, Chen LK, Fielding RA, Martin FC, Michel JP, Sieber C, Stout JR, Studenski SA, Vellas B, Woo J, Zamboni M, Cederholm T. Prevalence of and interventions for sarcopenia in ageing adults: a systematic review. Report of the International Sarcopenia Initiative (EWGSOP and IWGS). Age Ageing. 2014 Nov;43(6):748-59. doi: 10.1093/ageing/afu115. Epub 2014 Sep 21. PMID 25241753
- [Background] Morgan PT, Harris DO, Marshall RN, Quinlan JI, Edwards SJ, Allen SL, Breen L. Protein Source and Quality for Skeletal Muscle Anabolism in Young and Older Adults: A Systematic Review and Meta-Analysis. J Nutr. 2021 Jul 1;151(7):1901-1920. doi: 10.1093/jn/nxab055. PMID 33851213
- [Background] Gross DC, Cheever CR, Batsis JA. Understanding the development of sarcopenic obesity. Expert Rev Endocrinol Metab. 2023 Sep-Nov;18(6):469-488. doi: 10.1080/17446651.2023.2267672. Epub 2023 Nov 28. PMID 37840295
- [Background] Ferrucci L, de Cabo R, Knuth ND, Studenski S. Of Greek heroes, wiggling worms, mighty mice, and old body builders. J Gerontol A Biol Sci Med Sci. 2012 Jan;67(1):13-6. doi: 10.1093/gerona/glr046. Epub 2011 Nov 23. No abstract available. PMID 22113943
- [Background] Roubenoff R. Origins and clinical relevance of sarcopenia. Can J Appl Physiol. 2001 Feb;26(1):78-89. doi: 10.1139/h01-006. English, French. PMID 11291626
- [Background] Rosenberg IH. Sarcopenia: origins and clinical relevance. Clin Geriatr Med. 2011 Aug;27(3):337-9. doi: 10.1016/j.cger.2011.03.003. Epub 2011 Jun 8. PMID 21824550